CLINICAL TRIAL: NCT00677339
Title: Phase 3 Trial of Oral L-arginine and / or Vitamin D as Adjunctive Therapies in Pulmonary Tuberculosis in Papua Province, Indonesia.
Brief Title: L-arginine and Vitamin D Adjunctive Therapy in Pulmonary Tuberculosis (TB)
Acronym: AVDAPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other); Australian National University (Other)
Responsible Party: Principal Investigator, Dr Anna Ralph, Global and Tropical Health, Menzies School of Health Research
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVDAPT 1
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Smear Positive Pulmonary Tuberculosis
Keywords: Tuberculosis; Adjunctive therapy; L-arginine; Nitric oxide; Vitamin D
MeSH Terms: conditions — Tuberculosis | interventions — Arginine; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Active L-arginine plus active vitamin D
  Interventions: Drug: L-arginine; Drug: Vitamin D
- 2 (Active Comparator): Placebo L-arginine plus active Vitamin D
  Interventions: Drug: Vitamin D; Drug: Placebo L-arginine
- 3 (Active Comparator): Active L-arginine plus placebo vitamin D
  Interventions: Drug: L-arginine; Drug: Placebo Vitamin D
- 4 (Placebo Comparator): placebo L-arginine plus placebo vitamin D
  Interventions: Drug: Placebo L-arginine; Drug: Placebo Vitamin D

INTERVENTIONS:
Drug: L-arginine — L-arginine 6g orally daily
  Other Names: Argimax
  Arms: 1; 3
Drug: Vitamin D — Cholecalciferol 50000 IU once monthly orally
  Other Names: Calciferol Strong
  Arms: 1; 2
Drug: Placebo L-arginine — placebo L-arginine once daily
  Arms: 2; 4
Drug: Placebo Vitamin D — placebo vitamin D orally once monthly
  Arms: 3; 4

SUMMARY:
The purpose of this study is to determine whether adjunctive L-arginine and vitamin D can improve response to standard short course TB therapy in people with newly diagnosed pulmonary TB.

DETAILED DESCRIPTION:
The two major pathways proposed to mediate macrophage mycobacterial killing in humans are the arginine-nitric oxide and Vitamin D-1,25 dihydroxyvitamin D pathways. Our aim is to determine if the key immunomodulatory agents L-arginine and vitamin D can improve the rapidity and magnitude of the microbiological and clinical response in pulmonary TB. We will test the following hypotheses in newly-diagnosed TB patients in Timika, Papua, Indonesia:

Our specific aims are to:

1. Determine whether supplementation with L-arginine and/or vitamin D is safe, and results in more rapid improvement in clinical, mycobacterial, immunological, radiological, physiological and functional measures of treatment outcome. We will randomise patients with pulmonary TB to receive, in addition to standard TB therapy, adjunctive arginine, vitamin D and / or placebo in a randomised, double-blind factorial 2x2 design. We will relate serial measurements of plasma concentrations of L-arginine and vitamin D, and immunological responses (pulmonary NO production, T cell function and phenotype) to measures of treatment outcome [mycobacterial (sputum smear clearance and culture conversion), physiological (spirometry), clinical (symptoms and weight), radiological (chest Xray) and functional (six-minute walk test, modified St George Respiratory Questionnaire)].
2. Determine whether pulmonary production of NO is inversely related to disease severity at presentation. Baseline and serial measures of NO production will be related to disease severity and the magnitude and rapidity of clinical response

ELIGIBILITY:
Inclusion Criteria:

* Adults >15 years with sputum smear positive pulmonary TB
* New cases only
* Agree to continue treatment in Timika for the full six month course of treatment -Not pregnant
* Consent to enroll in the study.

Exclusion Criteria:

* hypercalcaemia (ionized calcium >1.32 mmol/L) identified at baseline
* taking arginine or vitamin D

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-06; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Proportion of pulmonary TB patients who are culture negative at 1 month | 1 month
Difference in improvement in composite clinical endpoint comprising weight, cough clearance and FEV1 at 2 months. | 2 months

SECONDARY OUTCOMES:
Change in plasma L-arginine concentration | week 0, 2, 4, 8, 24
Change in plasma 25(OH)D3 concentration | week 0, 2, 4, 8, 24
Death, clinical failure and default independently, and 'death or clinical failure or default'. | week 24
Hypercalcaemia | week 0, 2, 4, 8, 24
Gastrointestinal side effects | weekly to week 8 then at week 24
Sputum smear conversion time | weekly to week 8 then at week 24
Radiological improvement (percentage lung involvement on CXR at 2 months). | week 0, 2, 4, 8, 24
Cough clearance | weekly to week 8 then at week 24
Difference in improvement in percent predicted FEV1 at 2 and 6 months. | weeks 0, 4, 8, 24
Weight gain | weekly to week 8 then at week 24
Immunological improvement (exhaled NO) | week 0, 2, 4, 8, 24
Immunological improvement (T cell CD3ζ expression and T cell function) | week 0, 2, 4, 24
Functional improvement measured using six minute walk test | week 0, 4, 8, 24
Quality of life assessment using modified St George Respiratory Questionnaire. | weeks 0, 4, 8, 24
Primary end points stratified by HIV status. | weekly to week 8 then at week 24
Primary end points stratified by baseline vitamin D and L-arginine status. | weekly to week 8 then week 24
Primary end points stratified by ethnicity (Papuan and non-Papuan patients). | weekly to week 8 then week 24

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas M Anstey, MBBS, Study Director — Menzies School of Helath Research; Anna P Ralph, MBBS, Principal Investigator — Australian National University, Canberra, Australia; Franciscus Thio, MPPM, Principal Investigator — District Ministry of Health, Timika; Peter Morris, MBBS, Principal Investigator — Menzies School of Health Research, Northern Territory, Australia; Enny Kenangalem, MD, Principal Investigator — Papuan Community Health and Development Foundation; Jeanne R Poespoprodjo, MD, Principal Investigator — Mimika District Health Authority; Richard N Price, MD, Principal Investigator — Menzies School of Health Research; Tonia Woodberry, PhD, Principal Investigator — Menzies School of Health Research; Paul M Kelly, MBBS, Principal Investigator — Australian Capital Territory Department of Health; Emiliana Tjitra, MD, PhD, Principal Investigator — National Institute of Health Research and Development, Ministry of Health Republic of Indonesia; Sandjaja Sandjaja, PhD, Principal Investigator — National Institute of Health Research and Development, Ministry of Health Republic of Indonesia; Dina B Lolong, MD, Principal Investigator — National Institute of Health Research and Development; Mark Chatfield, PhD, Principal Investigator — National Health and Medical Research Council (Australia) Clinical Trials Centre; Ivan Bastian, MBBS, Principal Investigator — Institute of Medical and Veterinary Pathology, South Australia
Locations (1):
- Timika Tuberculosis Clinic and Community Hospital, Timika, Papua Province, Indonesia

REFERENCES:
- [Derived] Ralph AP, Waramori G, Pontororing GJ, Kenangalem E, Wiguna A, Tjitra E, Sandjaja, Lolong DB, Yeo TW, Chatfield MD, Soemanto RK, Bastian I, Lumb R, Maguire GP, Eisman J, Price RN, Morris PS, Kelly PM, Anstey NM. L-arginine and vitamin D adjunctive therapies in pulmonary tuberculosis: a randomised, double-blind, placebo-controlled trial. PLoS One. 2013 Aug 14;8(8):e70032. doi: 10.1371/journal.pone.0070032. eCollection 2013. PMID 23967066